CLINICAL TRIAL: NCT03469817
Title: Maveric Magnetic Resonance Imaging Used to Study Detailed Bone Apposition and Fixation of the Stryker Trident II Tritanium System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-1570
Record Dates: First submitted 2018-02-09; First posted 2018-03-19 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hip Pain
Keywords: Bone apposition; Stryker; MRI; Trident II; Total Hip Replacement

STUDY DESIGN:
Intervention Model Description: 1 control group who have had been implanted with a Trident cup and have already had MRIs taken at their one year post-operative visit. This group's MRI's will be compared with MRI's from Tridend II patients who have had MRI's at 1 year post-operative visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients who have undergone THR with Trident Cup (No Intervention): Patients who have had THR with Trident Cups and have previously had an MRI taken at the Hospital for Special Surgery at 1 year post-op.
- Patients who have undergone THR with Trident II Cup (Other): Patients who have had THR with Trident II Cups and will have an MRI taken at their one year post-operative visit.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Patients who are part of "Arm 2" will undergo an MRI at their 1 year post-operative visit.
  Arms: Patients who have undergone THR with Trident II Cup

SUMMARY:
The study aims to describe bone apposition and fixation of the Trident and Trident II Tritatnium acetabular system in patients 1 year status post total hip replacement. We will be studying this by comparing magnetic resonance imaging (MRI)s taken 1 year s/p total hip replacement with a Trident II cup with MRI's taken of patients with the Trident Cup who had MRIs done at 1 year post-op.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had a primary total hip replacement with a Stryker Trident II acetabular cup that have one year or more follow up.
2. Patients that are willing able able to have an MRI at their one year follow up visit.
3. Patients entered into the CORRe database (our HSS institutional joint replacement registry).

Exclusion Criteria:

1. Patients who have not been consented as part of the CORRe database.
2. Patients who are unable or refuse to have an MRI at their 1 year follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Comparison of bone apposition and fixation in patients with the Trident II Tritanium hip system with bone apposition and fixation in patients with Trident cups. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No